CLINICAL TRIAL: NCT03001869
Title: The Safety and Efficacy of 68Ga-HBED-CC-PSMA PET/CT in Prostate Cancer
Brief Title: 68Ga-PSMA PET/CT in Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephan Probst, MD, Chief of Nuclear Medicine, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-293
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-PSMA PET/CT (Experimental): 68Ga-HBED-CC-PSMA PET/CT
  Interventions: Drug: 68Ga-HBED-CC-PSMA PET/CT

INTERVENTIONS:
Drug: 68Ga-HBED-CC-PSMA PET/CT — 68Ga-HBED-CC-PSMA PET/CT Scan
  Other Names: 68Ga-PSMA-11

SUMMARY:
The objectives of this study are to replicate the safety and efficacy of 68Ga-PSMA PET/CT and as a diagnostic and decision making tool in the management prostate cancer patients.The primary endpoints of the study are the incidence of adverse events (AE) in the study population up to 7 days following the scan, and the sensitivity and specificity of 68Ga-PSMA PET/CT vs CT on a per-patient and per-lesion basis.

DETAILED DESCRIPTION:
Positron emission tomography / computer tomography (PET/CT) is a nuclear medicine diagnostic imaging procedure based on the measurement of positron emission from radiolabeled tracer molecules in vivo. A radiotracer in use today is 68Ga-HBED-CC-PSMA (DKFZ-11) - hereinafter abbreviated 68Ga-PSMA - which is a radiolabeled urea-based ligand for prostate specific membrane antigen (PSMA) PET/CT. Imaging with 68Ga-PSMA PET is used to characterize and localize prostate cancer in humans in vivo. There is extensive data in the literature showing the value of 68Ga-PSMA PET/CT imaging in accurately staging and restaging prostate cancer. The objectives of this study are to replicate the safety and efficacy of 68Ga-PSMA PET/CT and to establish our ability to reproduce results from the literature using 68Ga-PSMA PET/CT as a diagnostic and decision making tool in the management prostate cancer patients. During the study eligible prostate cancer patients will undergo one 68Ga-PSMA PET/CT. The primary endpoints of the study are the incidence of adverse events (AE) in the study population up to 7 days following the scan, and the sensitivity and specificity of 68Ga-PSMA PET/CT vs CT on a per-patient and per-lesion basis.

ELIGIBILITY:
Global Inclusion Criteria:

* Resident of Canada
* Male sex
* Age 18 years or older
* Previously diagnosed with prostate cancer, under referring physician's care
* ECOG performance status 0 - 3, inclusive
* Able to understand and provide written informed consent
* Able to tolerate the physical/logistical requirements of a PET/CT scan including lying supine (or prone) for up to 40 minutes and tolerating intravenous cannulation

Global Exclusion Criteria:

* Patients who are medically unstable (e.g. acute cardiac or respiratory distress or hypotensive)
* Patients who exceed the safe weight limit of the PET/CT bed (usually approximately 400 lbs.) or who cannot fit through the PET/CT bore (usually approximately 70 cm diameter)
* Patients with unmanageable claustrophobia

Clinical Indication Criteria Subgroups:

* BCR: Biochemical recurrence as defined by serum PSA > 0.1 ng/ml following either radical prostatectomy or curative-intent radiotherapy or other prostate-ablative definitive management
* HRS: Staging of high risk patients as defined by any one of the following:

  * Gleason score > 7
  * Serum PSA > 10 ng/ml
  * T stage of T3 or greater on TNM staging
  * Equivocal conventional staging such as CT, MRI or bone scan
  * Clinical suspicion of advance stage disease (e.g. bone pain)

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Safety of Ga68-PSMA PET/CT imaging as measured by the incidence of adverse events (AE) | 7 days
Efficacy of Ga68-PSMA PET/CT imaging as measured by sensitivity and specificity vs CT on a per patient basis as compared to standard of truth | 12 months
Efficacy of Ga68-PSMA PET/CT imaging as measured by sensitivity and specificity vs CT on a per lesion basis as compared to standard of truth | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided